CLINICAL TRIAL: NCT04551547
Title: A Randomized, Double-Blinded, Placebo-Controlled, Phase Ⅰ/Ⅱ Clinical Trial, to Evaluate the Safety and Immunogenicity of the SARS-CoV-2 Inactivated Vaccine (Vero Cell) in Healthy Population Aged 3-17 Years
Brief Title: Safety and Immunogenicity Study of Inactivated Vaccine for Prevention of COVID-19
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sinovac Research and Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-nCOV-1003
Record Dates: First submitted 2020-09-15; First posted 2020-09-16 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2021-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Vaccine-low dosage (Experimental): low dosage inactivated SARS-CoV-2 vaccine
  Interventions: Biological: Two doses of low dosage inactivated SARS-CoV-2 vaccine at the schedule of day 0,28
- Experimental Vaccine-medium dosage (Experimental): medium dosage inactivated SARS-CoV-2 vaccine
  Interventions: Biological: Two doses of medium dosage inactivated SARS-CoV-2 vaccine at the schedule of day 0,28
- Placebo (Placebo Comparator): No active ingredient in the placebo
  Interventions: Other: Two doses of placebo at the schedule of day 0,28

INTERVENTIONS:
Biological: Two doses of low dosage inactivated SARS-CoV-2 vaccine at the schedule of day 0,28 — The inactivated SARS-CoV-2 vaccine was manufactured by Sinovac Research & Development Co., Ltd., with a antigen content of 300SU/0.5ml
  Arms: Experimental Vaccine-low dosage
Biological: Two doses of medium dosage inactivated SARS-CoV-2 vaccine at the schedule of day 0,28 — The inactivated SARS-CoV-2 vaccine was manufactured by Sinovac Research & Development Co., Ltd., with a antigen content of 600SU/0.5ml
  Arms: Experimental Vaccine-medium dosage
Other: Two doses of placebo at the schedule of day 0,28 — The placebo contains no active ingredient and manufactured by Sinovac Research & Development Co., Ltd.
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blinded, and placebo controlled phase 1&2 clinical trial of the SARS-CoV-2 inactivated vaccine manufactured by Sinovac Research & Development Co., Ltd. The purpose of this study is to evaluate the safety and immunogenicity of the experimental vaccine in healthy children and adolescents aged 3-17 years

DETAILED DESCRIPTION:
This study is a randomized, double-blinded, single-center, placebo-controlled phase 1&2 clinical trial in children and adolescents aged 3-17 years. The experimental vaccine and placebo were both manufactured by Sinovac Research & Development Co., Ltd. A total of 552 subjects will be enrolled, with 72 at phase 1, and 480 at phase 2. Subjects will be assigned to receive two doses of different dosage of experimental vaccine or placebo on the schedule of day 0,28. Subjects in Phase receive the second dose 10 months or 12 months after the second dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children and adolescents aged 3-17 years;
* The subject and/or guardian can understand and voluntarily sign the informed consent form (double sign required for 8-17 years old);
* Proven legal identity.

Exclusion Criteria:

* Travel history / residence history of communities with case reports within 14 days;
* History of contact with a SARS-CoV-2 infection (positive in nucleic acid test) within 14 days;
* Have contacted patients with fever or respiratory symptoms from communities with case reports within 14 days;
* Two or more cases of fever and / or respiratory symptoms in a small contact area of volunteers, such as home, office etc. within 14 days;
* History of SARS-CoV-2 infection;
* History of asthma, history of allergy to the vaccine or vaccine components, or serious adverse reactions to the vaccine, such as urticaria, dyspnea, and angioedema;
* Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.;
* Autoimmune disease or immunodeficiency / immunosuppression;
* Severe chronic diseases, severe cardiovascular diseases, hypertension and diabetes that cannot be controlled by drugs, liver or kidney diseases, malignant tumors, etc.;
* Severe neurological disease (epilepsy, convulsions or convulsions) or mental illness;
* Thyroid disease or history of thyroidectomy, spleenlessness, functional spleenlessness, spleenlessness or splenectomy resulting from any condition;
* Diagnosed abnormal blood coagulation function (eg, lack of blood coagulation factors, blood coagulopathy, abnormal platelets) or obvious bruising or blood coagulation;
* Immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids (excluding allergic rhinitis corticosteroid spray therapy, acute noncomplicated dermatitis superficial corticosteroid therapy) in the past 6 months;
* Physical examination has clinically significant abnormal hematology and biochemistry laboratory test results that exceed the reference value range (only applicable to phase I clinical trials):

  1. Blood routine test: white blood cell count, hemoglobin, platelet count;
  2. Detection of blood biochemical indicators: alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin (TBIL), creatinine (CR), fasting blood glucose;
  3. Urine routine index: urine protein (PRO);
* History of alcohol or drug abuse;
* Receipt of blood products within in the past 3 months;
* Receipt of other investigational drugs in the past 30 days;
* Receipt of attenuated live vaccines in the past 14 days;
* Receipt of inactivated or subunit vaccines in the past 7 days;
* Acute diseases or acute exacerbation of chronic diseases in the past 7 days;
* Axillary temperature >37.0°C;
* Already pregnant (including a positive urine pregnancy test) or are breastfeeding, planning to get pregnant within 3 months;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 552 (Actual)
Dates: Start 2020-10-31 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
Safety index-incidence of adverse reactions | Day 0-28 after each dose vaccination
  Incidence of adverse reactions after each dose vaccination.
Immunogenicity index-seroconversion rates of neutralizing antibody | The 28th day after the second dose vaccination
  Neutralizing antibody assay will be performed using the micro-neutralization method. Seroconversion will be defined as a change from seronegative (<1:8) to seropositive (≥1:8), or ≥4 fold increase from baseline.

SECONDARY OUTCOMES:
Safety index-incidence of serious adverse events | From the beginning of the vaccination to 12 months after the second dose vaccination
  SAE will be collected throughout the clinical trial.
Immunogenicity index-seropositive rates of neutralizing antibody | The 28th day after each dose vaccination and the 12 month after the second dose vaccination
  Neutralizing antibody assay will be performed using the micro-neutralization method, and subjects with a antibody titer ≥1:8 will defined as seropositive.
Immunogenicity index-geometric mean titer (GMT) of neutralizing antibody | The 28th day after each dose vaccination and the 12 month after the second dose vaccination
  Neutralizing antibody assay will be performed using the micro-neutralization method.
Immunogenicity index-geometric mean ratio (GMR) of neutralizing antibody | The 28th day after each dose vaccination and the 12 month after the second dose vaccination
  Neutralizing antibody assay will be performed using the micro-neutralization method. Ratio of post-vaccination titer divided by baseline titer will be calculated.
Safety index-Incidence rate of adverse reactions | Within 7 days after each dose vaccination
  Incidence rate of adverse reactions within 7 days after each dose vaccination
Safety index-Incidence of abnormal laboratory index | On the 3th day after each dose of vaccination in phase Ⅰ
  Incidence of abnormal laboratory index (blood routine test, blood chemistry test, and urine routine test) on the 3th day after each dose of vaccination in phase Ⅰ
Safety index-Incidence rate of AESIs | From the beginning of the vaccination to 12 months after the last dose vaccination
  Incidence rate of SAEs and AESIs from the beginning of the vaccination to 12 months after the last dose vaccination
Immunogenicity index- GMI of neutralizing antibody | 28 days after the second dose vaccination
  GMI of neutralizing antibodies 28 days after the second dose vaccination
Immunogenicity index-the seroconversion rate | 28 days after the first dose vaccination in phase Ⅰ
  The seroconversion rate 28 days after the first dose vaccination in phase Ⅰ
Immunogenicity index-the seropositive rate | 28 days after the first dose vaccination in phase Ⅰ
  Seropositive rate 28 days after the first dose vaccination in phase Ⅰ
Immunogenicity index-the GMT | 28 days after the first dose vaccination in phase Ⅰ
  The GMT 28 days after the first dose vaccination in phase Ⅰ
Immunogenicity index-the GMI | 28 days after the first dose vaccination in phase Ⅰ
  The GMI 28 days after the first dose vaccination in phase Ⅰ

OTHER OUTCOMES:
Phase Ⅰ: The seropositive rate of neutralizing antibody | 6 months and 12 months after the second dose vaccination
  The seropositive rate of neutralizing antibody against live SARS-CoV-2 6 months and 12 months after the second dose vaccination
Phase Ⅰ:The GMT of neutralizing antibody | 6 months and 12 months after the second dose vaccination.
  The GMT of neutralizing antibody against live SARS-CoV-2 6 months and 12 months after the second dose vaccination.
Phase Ⅱ: The seropositive rate of neutralizing antibody | 3 months, 6 months, 9 months and 12 months after the second dose vaccination
  The seropositive rate of neutralizing antibody against live SARS-CoV-2 3 months, 6 months, 9 months and 12 months after the second dose vaccination
Phase Ⅱ: The GMT of neutralizing antibody | 3 months, 6 months, 9 months and 12 months after the second dose vaccination.
  The GMT of neutralizing antibody against live SARS-CoV-2 3 months, 6 months, 9 months and 12 months after the second dose vaccination.
Phase Ⅱ: The seropositive rate | 28 days after the booster dose
  The seropositive rate of neutralizing antibody against Prototype SARS-CoV-2 and Omicron strain 28 days after the booster dose
Phase Ⅱ: The GMT | 28 days after the booster dose
  The GMT of neutralizing antibody against Prototype SARS-CoV-2 and Omicron strain 28 days after the booster dose
Phase Ⅱ: The GMI | 28 days after the booster dose
  The GMI of neutralizing antibody against Prototype SARS-CoV-2 and Omicron strain 28 days after the booster dose
Phase Ⅱ: the seropositive rate | 6 months and 12 months after the booster dose
  The seropositive rate of neutralizing antibody against Prototype SARS-CoV-2 and Omicron strain 6 months and 12 months after the booster dose.
Phase Ⅱ: the GMT | 6 months and 12 months after the booster dose
  The GMT of neutralizing antibody against Prototype SARS-CoV-2 and Omicron strain 6 months and 12 months after the booster dose.

CONTACTS AND LOCATIONS:
Overall Officials: Yuliang Zhao, Master, Principal Investigator — Hubei Provincial Center for Disease Control and Prevention
Locations (1):
- Zanhuang county Center for Disease Control and Prevention, Shijiazhuang, Hebei, China

REFERENCES:
- [Derived] Han B, Song Y, Li C, Yang W, Ma Q, Jiang Z, Li M, Lian X, Jiao W, Wang L, Shu Q, Wu Z, Zhao Y, Li Q, Gao Q. Safety, tolerability, and immunogenicity of an inactivated SARS-CoV-2 vaccine (CoronaVac) in healthy children and adolescents: a double-blind, randomised, controlled, phase 1/2 clinical trial. Lancet Infect Dis. 2021 Dec;21(12):1645-1653. doi: 10.1016/S1473-3099(21)00319-4. Epub 2021 Jun 28. PMID 34197764